CLINICAL TRIAL: NCT00333788
Title: Open Label Long Term Clinical Trial Evaluating Efficacy and Safety of Chronic Therapy With Certolizumab Pegol, a PEGylated Fab Fragment of Humanized Antibody to Tumor Necrosis Factor Alpha (TNF) in Patients Suffering From Crohn's Disease and Having Completed C87042 Study.
Brief Title: Follow-up to Welcome Study C87042 [NCT00308581] Examining Certolizumab Pegol (CDP870) in Subjects With Crohn's Disease
Acronym: Welcome2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C87046; 2006-001729-24 (EudraCT Number)
Expanded Access: NCT03559660 (No longer available)
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Results first posted 2011-07-12 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2011-08

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Certolizumab pegol; CDP870; Cimzia
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Certolizumab pegol 400 mg (Experimental): 400 mg subcutaneous injection of certolizumab pegol every 2 (Q2W) or 4 (Q4W) weeks
  Interventions: Biological: Certolizumab pegol (CDP870)

INTERVENTIONS:
Biological: Certolizumab pegol (CDP870) — 400 mg subcutaneous (sc) injection of Certolizumab pegol (CDP870) every 2 (Q2W) or 4 (Q4W) weeks
  Other Names: CDP870; Cimzia

SUMMARY:
The study will continue to assess the safety of certolizumab pegol (CDP870) as well as examine the evolution of long term efficacy in Crohn's disease patients who completed study C87042 [NCT00308581]. It will also assess the effect of subcutaneous CDP870 400 mg on direct cost parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients having completed study C87042 [NCT00308581] (previously treated with infliximab)

Exclusion Criteria:

* Subject withdraw from C87042 [NCT00308581] study
* Subject who received treatment other than certolizumab pegol and other than medications permitted in C87042 [NCT00308581] study
* Subjects from countries where certolizumab pegol is authorized in Crohn's disease treatment
* Female patients of childbearing age who are NOT practicing (in the Investigator's opinion) effective birth control. All female patients must test negative on a serum pregnancy test before study entry and negative on urine testing immediately before every certolizumab pegol administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2006-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (65):
- United States (19):
  - Gainesville, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Lincoln, Nebraska
  - New York, New York
  - Chapel Hill, North Carolina
  - Charleston, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Charleston, South Carolina
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - Seattle, Washington
- Austria (2):
  - Innsbruck
  - Vienna
- Belgium (7):
  - Bonheiden
  - Brussels
  - Genk
  - Ghent
  - Leuven
  - Liège
  - Roeselare
- Canada (5):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - London, Ontario
  - Toronto, Ontario
  - Calgary
- France (5):
  - Clichy
  - Lille
  - Nice
  - Paris
  - Pessac
- Germany (8):
  - Berlin
  - Hamburg
  - Herne
  - Kiel
  - Leipzig
  - Minden
  - Munich
  - München
- Italy (6):
  - Bologna
  - Milan
  - Padua
  - Palermo
  - Roma
  - Torino
- Netherlands (2):
  - Eindhoven
  - Heerlen
- Spain (5):
  - Barcelona
  - Madrid
  - Santiago de Compostela
  - Seville
  - Valencia
- Stockholm, Sweden
- Switzerland (2):
  - Bern
  - Lausanne
- United Kingdom (3):
  - Bristol
  - London
  - Oxford

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started in October 2006, with recruitment in the United States, Austria, Belgium, Canada, France, Germany, Italy, Spain, Sweden, Switzerland, the United Kingdom and the Netherlands. This study completed in April 2010.
Pre-assignment Details: The summary of Participant Flow is based on the All Subjects Population.
Period: Overall Study
Arm/Group | Certolizumab Pegol 400 mg
Started | 233 (Participant flow based on All Subjects population; Baseline characteristics based on ITT population.)
Completed | 71
Not Completed | 162
Not completed — Adverse Event | 44
Not completed — Lack of Efficacy | 80
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 24
Not completed — Other: Non-compliance | 2
Not completed — Other: Moved | 2
Not completed — Other: Recurrent squamaous cell cancer | 1
Not completed — Other: Investigator decision | 1
Not completed — Other: Quality of life concern | 1
Not completed — Other: Sponsor decision | 1
Not completed — Other: Subject in need of an Entocort | 1
Not completed — Other: Medical monitor decision | 1
Not completed — Other: Physician decision | 1
Not completed — Other: Signed consent for another study | 1

BASELINE CHARACTERISTICS:
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
Age, Categorical [Count of Participants; unit: Participants] — Baseline characteristics are based on the ITT population; Participant flow is based on the All Subjects population.
  Participants
    <=18 years | 1
    Between 18 and 65 years | 224
    >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline characteristics are based on the ITT population; Participant flow is based on the All Subjects population.
  years | 31.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics are based on the ITT population; Participant flow is based on the All Subjects population.
  Participants
    Female | 146
    Male | 83
Region of Enrollment [Number; unit: participants] — Baseline characteristics are based on the ITT population; Participant flow is based on the All Subjects population.
  participants
    France | 20
    United States | 70
    Canada | 20
    Spain | 6
    Belgium | 30
    Austria | 8
    Netherlands | 2
    Germany | 34
    United Kingdom | 9
    Switzerland | 4
    Italy | 24
    Sweden | 2

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of at Least One Study-emergent Adverse Event During the Study (Maximum 164 Weeks)
Description: Study-emergent adverse events are defined as treatment-emergent adverse events with an onset date on or after the first study drug administration date of this study but not later than 12 weeks (84 days) after last injection.
  Results are presented as the percentage of subjects with at least one treatment-emergent adverse event during this study.
Time Frame: Maximum 164 weeks
Population: Of the 233 subjects in the study, 229 are in the Intent to Treat (ITT) population and are included in this analysis. Note that the ITT population is the same as the Safety Set (SS) population.
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
percentage of participants | 92.6

2. Secondary Outcome: Maintenance of Response at Last Visit [Up to the Maximum Study Duration Observed in the Study (Week 154) or the Withdrawal Visit for Premature Withdrawals] Among the Subjects in Clinical Response at Baseline of This Study (Week 26 of Study C87042).
Description: Clinical response is defined as at least a 100 point decrease from Baseline of study C87042 (NCT00308581) in Crohn's Disease Activity Index (CDAI).
  Subjects maintained their clinical response at Last Visit if they did not meet criteria for loss of response [CDAI score >150 points and a minimum increase in CDAI of 70 points versus Baseline of study C87042 (NCT00308581)] at 2 consecutive visits.
  A CDAI score of 150 or below indicates remission and a score above 450 indicates extremely severe disease.
  Results are presented as the percentage of subjects maintaining response at Last visit.
Time Frame: Baseline (corresponding to Week 26 of study C87042 (NCT00308581) and Last Visit [Up to the maximum study duration observed in the study (Week 154) or the Withdrawal Visit for Premature Withdrawals]
Population: Of the 233 subjects in the study, 166 are in the Intent to Treat (ITT) population and were in clinical response at Baseline of this study, and are included in this analysis. Note that the ITT population is the same as the Safety Set (SS) population.
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 166
percentage of participants | 61.8

3. Secondary Outcome: Clinical Response at Last Visit [Up to the Maximum Study Duration Observed in the Study (Week 154) or the Withdrawal Visit for Premature Withdrawals]
Description: Clinical response is defined as at least a 100 point decrease from Baseline of study C87042 (NCT00308581) in Crohn's Disease Activity Index (CDAI).
  CDAI is used to quantify the symptoms of Crohn's disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease.
  Results are presented as the percentage of subjects achieving clinical response at Last visit.
Time Frame: Baseline of study C87042 (NCT00308581) and Last Visit [Up to the maximum study duration observed in the study (Week 154) or the Withdrawal Visit for Premature Withdrawals]
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
percentage of participants | 53.3

4. Secondary Outcome: Remission at Last Visit [Up to the Maximum Study Duration Observed in the Study (Week 154) or the Withdrawal Visit for Premature Withdrawals]
Description: Remission is defined as a Crohn's Disease Activity Index (CDAI) score ≤ 150 points
  CDAI is used to quantify the symptoms of Crohn's disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease.
  Results are presented as the percentage of subjects in remission at Last visit.
Time Frame: Last Visit [Up to the maximum study duration observed in the study (Week 154) or the Withdrawal Visit for Premature Withdrawals]
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
percentage of participants | 40.6

5. Secondary Outcome: Change From Baseline of Study C87042 (NCT00308581) in Crohn's Disease Activity Index (CDAI) at Last Visit [Up to the Maximum Study Duration Observed in the Study (Week 154) or the Withdrawal Visit for Premature Withdrawals]
Description: CDAI is used to quantify the symptoms of Crohn's disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease.
Time Frame: as for outcome 3
Population: Of the 233 subjects in the study, 215 are in the Intent to Treat (ITT) population with Crohn's Disease Activity Index (CDAI) scores at Baseline and Last/Withdrawal visits and are included in this analysis. Note that the ITT population is the same as the Safety Set (SS) population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 215
score on a scale | -121.52 (99.61)

6. Secondary Outcome: Time to Loss of Response After Baseline of Study C87042 (NCT00308581) on Subjects Who Were in Clinical Response at Baseline of This Study
Description: Clinical response at Baseline of this study of at least a 100 point decrease from Baseline of study C87042 in Crohn's Disease Activity Index (CDAI)
  Loss of response = both a CDAI score >150 points and a minimum increase in CDAI of 70 points versus Baseline (Week 26 of study C87042) as confirmed at 2 consecutive visits. Subjects losing response will be considered as having the event on the date of the first visit where response was lost. Subjects who discontinued the study without having lost response will be censored on the date of discontinuation (i.e. date of last visit performed).
Time Frame: Maximum 154 weeks
Population: Of the 233 subjects in the study 153 are in the Modified Intent to Treat (MITT) population and are responders at Baseline of this study and are in this analysis. The MITT population includes subjects that are in the ITT population that were correctly randomized at Week 6 of study C87042 (NCT00308581).
Measure: Median (Full Range); unit: days
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 153
days | 169.5 (274.1) [85 to 814]

7. Secondary Outcome: Occurrence of at Least 1 Hospital Stay During the Treatment Period
Description: The Treatment Period is defined from the first administration of study drug in C87046 to the last/withdrawal study drug administration visit.
  Results are presented as the percentage of subjects with at least 1 hospital stay during the treatment period.
Time Frame: Maximum 152 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
percentage of participants | 21.4 (0.730)

8. Secondary Outcome: Occurrence of at Least 1 Hospital Stay During the Follow-Up Period
Description: Follow-up period starts the day after the last injection up to 84 days after last injection.
  Results are presented as the percentage of subjects with at least 1 hospital stay during the follow-up period.
Time Frame: Maximum 12 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
percentage of participants | 21.8 (0.578)

9. Secondary Outcome: Occurrence of at Least 1 Hospital Stay During the During the Overall Period
Description: Overall period corresponds to both treatment and follow-up periods in C87046.
  Results are presented as the percentage of subjects with at least 1 hospital stay during the overall period.
Time Frame: Maximum 164 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
percentage of participants | 37.6 (0.953)

10. Secondary Outcome: Length of Hospital Stays During the Treatment Period
Description: The Treatment Period is defined from the first administration of study drug in C87046 to the last/withdrawal study drug administration visit.
Time Frame: Maximum 152 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
days | 1.838 (5.785)

11. Secondary Outcome: Length of Hospital Stays During the Follow-Up Period
Description: Follow-up period starts the day after the last injection up to 84 days after last injection.
Time Frame: Maximum 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
days | 2.782 (7.743)

12. Secondary Outcome: Length of Hospital Stays During the Overall Period
Description: Overall period corresponds to both treatment and follow-up periods in C87046.
Time Frame: Maximum 164 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
days | 4.620 (9.704)

13. Secondary Outcome: Occurrence of at Least 1 Emergency Room Visit During the Treatment Period
Description: The Treatment Period is defined from the first administration of study drug in C87046 to the last/withdrawal study drug administration visit.
  Results are presented as the percentage of subjects with at least 1 emergency room visit during the treatment period.
Time Frame: Maximum 152 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
percentage of participants | 13.1 (0.413)

14. Secondary Outcome: Occurrence of at Least 1 Emergency Room Visit During the Follow-Up Period
Description: Follow-up period starts the day after the last injection up to 84 days after last injection.
  Results are presented as the percentage of subjects with at least 1 emergency room visit during the follow-up period.
Time Frame: Maximum 12 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
percentage of participants | 6.1 (0.265)

15. Secondary Outcome: Occurrence of at Least 1 Emergency Room Visit During the Overall Period
Description: Overall period corresponds to both treatment and follow-up periods in C87046.
  Results are presented as the percentage of subjects with at least 1 emergency room visit during the overall period.
Time Frame: Maximum 164 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
percentage of participants | 19.2 (0.471)

16. Secondary Outcome: Occurrence of at Least One Concomitant Medication Potentially Influencing Crohn's Disease During the Treatment Period
Description: The Treatment Period is defined from the first administration of study drug in C87046 to the last/withdrawal study drug administration visit.
  Medication categories are anti tumor necrosis factor (anti-TNFs), immunosuppressants, corticosteroids, 5 aminosalicylic acid (5-ASA) and antibiotics.
  Results are presented as the percentage of subjects with at least 1 concomitant medication potentially influencing Crohn's disease during the treatment period.
Time Frame: Maximum 152 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
percentage of participants
  Anti tumor necrosis factor (Anti-TNF) | 0.4 (0.066)
  Immunosuppressants | 3.9 (0.195)
  Corticosteroids | 24.0 (0.733)
  5- Aminosalicylic Acid (5-ASA) | 5.2 (0.356)
  Antibiotics | 55.5 (2.889)

17. Secondary Outcome: Occurrence of at Least One Concomitant Medication Potentially Influencing Crohn's Disease During the Follow-Up Period
Description: Follow-up period start the day after the last injection up to 84 days after last injection.
  Medication categories are anti tumor necrosis factor (anti-TNFs), immunosuppressants, corticosteroids, 5 aminosalicylic acid (5-ASA) and antibiotics.
  Results are presented as the percentage of subjects with at least 1 concomitant medication potentially influencing Crohn's disease during the follow-up period.
Time Frame: Maximum 12 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
percentage of participants
  Anti tumor necrosis factor (Anti-TNF) | 16.2 (0.702)
  Immunosuppresants | 5.2 (0.250)
  Corticosteroids | 15.3 (0.622)
  5- Aminosalicylic Acid (5-ASA) | 2.2 (0.185)
  Antibiotics | 14.0 (0.829)

18. Secondary Outcome: Occurrence of at Least One Concomitant Medication Potentially Influencing Crohn's Disease During the Overall Period
Description: Overall period corresponds to both treatment and follow-up periods in C87046.
  Medication categories are anti tumor necrosis factor (anti-TNFs), immunosuppressants, corticosteroids, 5 aminosalicylic acid (5-ASA) and antibiotics.
  Results are presented as the percentage of subjects with at least 1 concomitant medication potentially influencing Crohn's disease during the overall period.
Time Frame: Maximum 164 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
percentage of participants
  Anti tumor necrosis factor (Anti-TNF) | 16.2 (0.716)
  Immunosuppressants | 8.3 (0.337)
  Corticosteroids | 35.4 (0.986)
  5- Aminosalicylic Acid (5-ASA) | 7.0 (0.408)
  Antibiotics | 62.4 (2.974)

19. Secondary Outcome: Occurrence of at Least 1 General Concomitant Medication During the Treatment Period
Description: The Treatment Period is defined from the first administration of study drug in C87046 to the last/withdrawal study drug administration visit.
  Results are presented as the number of subjects who used at least 1 concomitant medication during the treatment period.
Time Frame: Maximum 152 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
participants | 185 (10.172)

20. Secondary Outcome: Occurrence of at Least 1 General Concomitant Medication During the Follow-Up Period
Description: Follow-up period start the day after the last injection up to 84 days after last injection.
  Results are presented as the number of subjects who used at least 1 concomitant medication during the follow-up period.
Time Frame: Maximum 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
participants | 71 (3.395)

21. Secondary Outcome: Occurrence of at Least 1 General Concomitant Medication During the Overall Period
Description: Overall period corresponds to both treatment and follow-up periods in C87046.
  Results are presented as the number of subjects who used at least 1 concomitant medication during the overall period.
Time Frame: Maximum 164 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
participants | 195 (10.948)

22. Secondary Outcome: Occurrence of at Least 1 Concurrent Medical Procedure During the Treatment Period.
Description: The Treatment Period is defined from the first administration of study drug in C87046 to the last/withdrawal study drug administration visit.
  Results are presented as the number of subjects who had at least 1 concurrent medical procedure during the treatment period.
Time Frame: Maximum 152 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
participants | 148 (4.656)

23. Secondary Outcome: Occurrence of at Least 1 Concurrent Medical Procedure During the Follow-Up Period
Description: Follow-up period start the day after the last injection up to 84 days after last injection.
  Results are presented as the number of subjects who had at least 1 concurrent medical procedure during the follow-up period.
Time Frame: Maximum 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
participants | 84

24. Secondary Outcome: Occurrence of at Least 1 Concurrent Medical Procedure During the Overall Period
Description: Overall period corresponds to both treatment and follow-up periods in C87046.
  Results are presented as the number of subjects who had at least 1 concurrent medical procedure during the overall period.
Time Frame: Maximum 164 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Certolizumab Pegol 400 mg
Number analyzed (Participants) | 229
participants | 173

ADVERSE EVENTS:
Time Frame: Maximum of 166 weeks
Description: Adverse Event reporting is based on the Safety population; Participant flow is based on the All Subjects population.
Arm/Group | Certolizumab Pegol 400 mg
Serious Adverse Events (participants affected / at risk) | 73/229
Other Adverse Events (participants affected / at risk) | 190/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol 400 mg (N=229)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (5)
Anal fistula (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Colonic stenosis (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 22 (23)
Faecal incontinence (Gastrointestinal disorders) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 1 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Hernial eventration (Gastrointestinal disorders) | 1 (1)
Ileal stenosis (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Intestinal stenosis (Gastrointestinal disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Rectal perforation (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Small intestinal stenosis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 3 (3)
Pyrexia (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Abdominal abscess (Infections and infestations) | 5 (5)
Abdominal wall abscess (Infections and infestations) | 1 (1)
Anal abscess (Infections and infestations) | 2 (2)
Breast abscess (Infections and infestations) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1)
Empyema (Infections and infestations) | 1 (1)
Fusobacterium infection (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2)
Infective tenosynovitis (Infections and infestations) | 1 (1)
Parotitis (Infections and infestations) | 1 (1)
Perianal abscess (Infections and infestations) | 5 (7)
Perineal abscess (Infections and infestations) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Rectal abscess (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 2 (3)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (2)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 2 (4)
Cerebral infarction (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Hyporeflexia (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Wallenberg syndrome (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol 400 mg (N=229)
Abdominal pain (Gastrointestinal disorders) | 45 (63)
Abdominal pain upper (Gastrointestinal disorders) | 18 (23)
Anal fissure (Gastrointestinal disorders) | 14 (16)
Constipation (Gastrointestinal disorders) | 14 (20)
Crohn's disease (Gastrointestinal disorders) | 41 (48)
Diarrhoea (Gastrointestinal disorders) | 33 (44)
Haematochezia (Gastrointestinal disorders) | 14 (16)
Nausea (Gastrointestinal disorders) | 23 (43)
Vomiting (Gastrointestinal disorders) | 24 (34)
Asthenia (General disorders) | 12 (15)
Fatigue (General disorders) | 21 (29)
Pyrexia (General disorders) | 47 (93)
Bronchitis (Infections and infestations) | 23 (33)
Gastroenteritis (Infections and infestations) | 16 (20)
Herpes simplex (Infections and infestations) | 24 (39)
Influenza (Infections and infestations) | 30 (35)
Nasopharyngitis (Infections and infestations) | 63 (117)
Sinusitis (Infections and infestations) | 23 (30)
Upper respiratory tract infection (Infections and infestations) | 12 (15)
Urinary tract infection (Infections and infestations) | 19 (31)
Arthralgia (Musculoskeletal and connective tissue disorders) | 44 (68)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (31)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (19)
Headache (Nervous system disorders) | 47 (80)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (31)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 21 (27)
Rash (Skin and subcutaneous tissue disorders) | 20 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.